CLINICAL TRIAL: NCT06145945
Title: A Randomized Controlled Study of the Effect of Intraperitoneal Ropivacaine on Visceral Pain After Laparoscopic Gastrectomy
Brief Title: Effect of Intraperitoneal Ropivacaine on Visceral Pain After Laparoscopic Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SanQing Jin (Other)
Responsible Party: Sponsor-Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023ZSLYEC-502
Record Dates: First submitted 2023-11-09; First posted 2023-11-24 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Laparoscopic Gastrectomy; Ropivacaine
Keywords: visceral pain
MeSH Terms: conditions — Visceral Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Experimental): 20ml 0.5% ropivacaine is sprayed intraperitoneally
  Interventions: Drug: 0.5% Ropivacaine
- Saline (Placebo Comparator): 20ml saline is sprayed intraperitoneally
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: 0.5% Ropivacaine — 20ml 0.5% ropivacaine is sprayed intraperitoneally
  Other Names: Ropivacaine
  Arms: Ropivacaine
Drug: Saline — 20ml saline is sprayed intraperitoneally
  Arms: Saline

SUMMARY:
Visceral pain is obvious and lasts for a long time in patients after laparoscopic gastrectomy.Relieving the visceral pain is of great significance for patients' postoperative emotional experience, functional recovery and reducing the formation of long-term chronic pain. However, there is no clear clinical consensus on relieving visceral pain by now, so effective clinical methods to relieve visceral pain need to be explored urgently.

Intraperitoneal spraying local anesthetics is a simple and inexpensive method, which has been proved to be safe and effective in randomized controlled trials and Meta-analysis of various types of surgery.However, its effect in clinical research is still controversial and many studies lack evaluation of postoperative recovery quality, so it has not been widely used in clinical practice.

This study aims to explore the effect of intraperitoneal spraying ropivacaine (long-acting amide local anesthetic) on visceral pain after laparoscopic gastrectomy, and to systematically evaluate its effect on the recovery of gastrointestinal function and the inflammatory factors (IL-6, TNF-α) in abdominal drainage fluid.

DETAILED DESCRIPTION:
Postoperative pain is a common adverse reaction after laparoscopic gastrectomy. Insufficient analgesia can cause severe stress response,affect the recovery of postoperative gastrointestinal function, increase the incidence of postoperative complications and prolong the length of hospital stay. Although laparoscopic surgery significantly reduces postoperative pain compared to traditional open surgery, the management of postoperative pain remains a challenge. Postoperative pain after laparoscopic surgery is mainly divided into three parts: incision pain(somatic pain component), deep abdominal pain (visceral pain component) and shoulder pain (referred pain component). In a prospective study, Blichfeldt-Eckhardt et al. found that visceral pain accumulated in the first week after surgery was identified as an independent risk factor for unexplained chronic pain at 12 months after surgery, and visceral pain was the only pain component that was independently and significantly associated with chronic unexplained pain at 12 months after surgery .

Visceral pain is generally defined as pain caused inside the body, but is usually caused by excessive contraction, stretching, or ischemia of the walls of internal organs . In contrast to pain signals originating from the skin,pain originating from the viscera is described as dull and diffuse, often poorly localized, and can be distant from its origin.Visceral pain is considered more unpleasant and frightening than somatic pain.

Therefore,relieving the visceral pain is of great significance for patients' postoperative emotional experience, functional recovery and reducing the formation of long-term chronic pain. However, there is no clear clinical consensus on relieving visceral pain by now, so effective clinical methods to relieve visceral pain need to be explored urgently.

Intraperitoneal spraying local anesthetics is a simple and inexpensive method, which has been proved to be a safe and effective way to reduce the use of opioid and postoperative pain score in randomized controlled trials and Meta-analysis of various surgical types such as laparoscopic cholecystectomy , laparoscopic appendectomy , laparoscopic gynecology and so on. Intraperitoneal spraying local anesthetics is a type of topical anesthesia.Local anesthetics produce local anesthesia by acting on nerve endings on the surface of the visceral organs.Visceral organs mainly transmit nociceptive signals through the vagus nerve and spinal nerve, among which the spinal nerve mainly transmits mechanical stimulation signals, while the vagus nerve mainly transmits chemical stimulation signals. Arman Kahokehr et al. found that intraperitoneal spraying local anesthetics during colectomy may reduce postoperative pain by blocking intra-abdominal vagus nerve signals. At the same time, it inhibits the corresponding neuroendocrine stress pathway, thus resulting in behavioral benefits. However, it does not separately evaluate the different pain components of patients after surgery.

At the same time,the effect of intraperitoneal spraying local anesthetics is still controversial and many studies lack evaluation of postoperative recovery quality,so this technique has not been widely used in clinical practice. Schipper IE et al. spray 20ml 2.5% bupivacaine into the abdominal cavity during laparoscopic gastric bypass surgery, and the test results indicated that the experimental group did not significantly reduce postoperative pain or opioid use, and the use of antiemetic drugs and the length of hospital stay were not significantly reduced.A review in 2021 included 85 clinical trials of intraperitoneal spraying local anesthetics during laparoscopic cholecystectomy, found that intraperitoneal spraying local anesthetics could reduce pain for up to 24 hours in patients undergoing laparoscopic cholecystectomy. However,none of these trials provided postoperation follow-up information and evaluation of postoperative recovery quality.

In this study, pain types are assessed independently to explore whether intraperitoneal spraying local anesthetics could reduce visceral pain by blocking splanchnic nerve afferents. This study will use ropivacaine, the most commonly used long-acting amide local anesthetic, which has low toxicity and an effective acting time of about 4-6 hours.This study set up multiple time points after surgery to evaluate the visceral pain and recovery quality of patients,in order to explore whether early postoperative pain control can slow down or block the formation of postoperative chronic pain, and systematically evaluate the effect of intraperitoneal spraying local anesthetics on the postoperative recovery quality of patients.In a meta-analysis Sparreboom CL et al. found that patients with postoperative anastomotic leakage had significantly higher levels of IL-6 and TNF-α in abdominal drainage fluid at 24h after surgery than those without anastomotic leakage, but this significant change was not observed in blood samples.Wiik et al. reported that inflammatory cytokines are more widely released into the abdominal cavity after abdominal surgery compared with systemic responses,which may be due to the secretion of these cytokines by lymphocytes and monocytes at the site of anastomotic leak.Inflammatory factors are not only related to postoperative anastomotic leakage, but also closely related to the occurrence and development of postoperative pain.Inflammatory stimulation or tissue damage stimulates a cytokine cascade that ultimately triggers the release of mediators that cause inflammatory pain. Immune cells release inflammatory factors such as IL-6 and TNF-α, and induce prostaglandin synthesis and enhance TRP and Nav channel activation through a series of signal transduction pathways, thus inducing inflammatory pain in vivo.Therefore, we plan to detect the inflammatory factors IL-6 and TNF-α in the abdominal drainage fluid at 24h after surgery,to explore the effect of Intraperitoneal spraying local anesthetics on the postoperative abdominal drainage fluid related inflammatory factors, and to evaluate its influence on the recovery of postoperative gastrointestinal function further.

The anesthesia induction protocol for this study includes intravenous titration administration of propofol at a rate of 0.5mg/kg/min, sufentanil 0.3ug/kg, and cisatracurium 0.2mg/kg. Anesthesia is maintained with propofol, remifentanil cisatracurium and sevoflurane to maintain the patient's blood pressure at ±20% of the basic blood pressure and BIS between 40 and 60. The first dose of analgesia and antiemetic (0.3ug/kg sufentanil + 5mg dezocine + 0.25mg palonosetron hydrochloride) is given half an hour before the end of surgery. Before closing the abdominal cavity after abdominal irrigation, 20ml of 0.5% ropivacaine or an equal volume of normal saline is uniformly sprayed onto the surgical area using an endoscopic instrument channel. After skin closure, 10ml of 0.5% ropivacaine is used for infiltration anesthesia at the incision site, and a venous analgesia pump is connected (3ug/kg sufentanil + dezocine 15mg+ palonosetron hydrochloride 0.5mg+NS 120ml). After the surgery, the patient is induced to spontaneous breathe and the tracheal tube will be removed, and then he is sent to the PACU for further observation. If the pain NRS score in the recovery room is greater than 4, a single injection of 5ug sufentanil will be administered until the NRS score is ≤4. When the patient achieve a Sterward score of 6 points, he will be returned to the ward.

Visceral pain is obvious and lasts for a long time in patients after laparoscopic gastrectomy. This study intends to include these patients in the study, and adopt ropivacaine, a local anesthetic with less cardiotoxicity and relatively long acting time,to provide further clinical data for the relief of postoperative visceral pain by intraperitoneal spraying local anesthetics.This study will also systematically evaluate the effect of intraperitoneal spraying local anesthetics on the postoperative recovery quality and the inflammatory factors in postoperative abdominal drainage fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. The American Society of Anesthesiologists(ASA) grade is I or II, and the heart function grade is 1-2;
3. Elective laparoscopic gastrectomy under general anesthesia

Exclusion Criteria:

1. Patients have severe heart, lung, liver, and kidney diseases (heart function grade>3 / respiratory failure / liver failure / renal failure)
2. BMI<18kg/m2 or >30kg/m2
3. Patients with chronic pain other than stomach pain and taking analgesics for a long time
4. Patients with history of allergy to local anesthetics
5. Patients with high risk of reflux and aspiration such as digestive obstruction
6. Patients who refuse to participate or don't sign or refuse to sign the informed consent form
7. Patients who are unable to communicate effectively
8. Patients participate in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
NRS scores of visceral pain | 24 hours after surgery
  NRS scores of visceral pain at 24 hours after surgery

SECONDARY OUTCOMES:
NRS scores of visceral pain | From surgery completion to the 30th day after surgery
  NRS scores of visceral pain at 0 hour,1 hour,6 hours,12 hours,the second day,the third day and the 30th day after surgery
NRS scores of incisional pain | From surgery completion to the 30th day after surgery
  NRS scores of incisional pain at 0 hour,1 hour,6 hours,12 hours,24 hours,the second day,the third day and the 30th day after surgery
NRS scores of referred pain | From surgery completion to the 30th day after surgery
  NRS scores of referred pain at 0 hour,1 hour,6 hours,12 hours,24 hours,the second day,the third day and the 30th day after surgery
Blood pressure(SBP,DBP,MAP) | From the period of anesthesia to the third day after surgery
  Relative change of blood pressure(SBP,DBP,MAP) at the time of entering the operating room,the beginning of anesthesia,the beginning of surgery and 0 hour,1 hour,6 hours,12 hours,24 hours,the second day,the third day after surgery
Heart rate | From the period of anesthesia to the third day after surgery
  Relative change of heart rate at the time of entering the operating room,the beginning of anesthesia,the beginning of surgery and 0 hour,1 hour,6 hours,12 hours,24 hours,the second day,the third day after surgery
Oxygen saturation | From the period of anesthesia to the third day after surgery
  Relative change of oxygen saturation at the time of entering the operating room,the beginning of anesthesia,the beginning of surgery and 0 hour,1 hour,6 hours,12 hours,24 hours,the second day,the third day after surgery
Additional analgesics in the ward | From surgery completion to the third day after surgery
  Use of additional analgesics in the ward
Nausea and vomiting | From surgery completion to the third day after surgery
  Whether nausea and vomiting, the frequency of vomiting
Use of intravenous analgesia pump | From surgery completion to the third day after surgery
  The total and effective pressing times of intravenous analgesia pump,total consumption of sufentanil
Serum C-reactive protein (CRP) concentration | One day before surgery and 24 hours after surgery
  Serum C-reactive protein (CRP) concentration
The level of blood glucose | One day before surgery and 24 hours after surgery
  The level of blood glucose
Interleukin-6(IL-6) | 24 hours after surgery
  IL-6 concentration in abdominal drainage fluid
Tumor necrosis factor-α(TNF-α) | 24 hours after surgery
  TNF-α concentration in abdominal drainage fluid
Postoperative recovery score using 15-item quality of recovery scoring system(QoR-15) | From the first day to the 30th day after surgery
  To evaluate the postoperative recovery using 15-item quality of recovery scoring system including emotional state,body comfort, psychological support, body independence and pain at the first day,the second day,the third day and the 30th day after surgery
Anal exhaust time | From surgery completion to first anal exhaust after surgery,assessed up to 7 days
  The time of first anal exhaust time after surgery
Sitting up time | From surgery completion to first sitting up after surgery,assessed up to 7 days
  The time of first sitting up time after surgery
Getting out of bed time | From surgery completion to first getting out of bed after surgery,assessed up to 7 days
  The time of first getting out of bed time after surgery
First drinking time after surgery | From surgery completion to first drinking after surgery,assessed up to 7 days
  First drinking time after surgery
First eating time after surgery | From surgery completion to first eating after surgery,assessed up to 7 days
  First eating time after surgery
Removal of stomach tube time | From surgery completion to removal of stomach tube,assessed up to 30 days
  Removal of stomach tube time
Removal of drainage tube time | From surgery completion to removal of drainage tube,assessed up to 30 days
  Removal of drainage tube time
Removal of indwelling urinary catheter time | From surgery completion to removal of indwelling urinary catheter,assessed up to 30 days
  Removal of indwelling urinary catheter time
Incidence of postoperative complications within 30 days after surgery | Within 30 days after surgery
  Incidence of intra-abdominal infection and anastomotic leakage within 30 days after surgery
Length of hospital stay after surgery | From surgery completion to actual hospital discharge, assessed up to 30 days
  Hospital stay time from operation completion to actual hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: SanQing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- SanQing Jin, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cha SM, Kang H, Baek CW, Jung YH, Koo GH, Kim BG, Choi YS, Cha SJ, Cha YJ. Peritrocal and intraperitoneal ropivacaine for laparoscopic cholecystectomy: a prospective, randomized, double-blind controlled trial. J Surg Res. 2012 Jun 15;175(2):251-8. doi: 10.1016/j.jss.2011.04.033. Epub 2011 May 17. PMID 21658722
- [Background] Blichfeldt-Eckhardt MR, Ording H, Andersen C, Licht PB, Toft P. Early visceral pain predicts chronic pain after laparoscopic cholecystectomy. Pain. 2014 Nov;155(11):2400-7. doi: 10.1016/j.pain.2014.09.019. Epub 2014 Sep 22. PMID 25250720
- [Background] Feng B, Guo T. Visceral pain from colon and rectum: the mechanotransduction and biomechanics. J Neural Transm (Vienna). 2020 Apr;127(4):415-429. doi: 10.1007/s00702-019-02088-8. Epub 2019 Oct 9. PMID 31598778
- [Background] Boezaart AP, Smith CR, Chembrovich S, Zasimovich Y, Server A, Morgan G, Theron A, Booysen K, Reina MA. Visceral versus somatic pain: an educational review of anatomy and clinical implications. Reg Anesth Pain Med. 2021 Jul;46(7):629-636. doi: 10.1136/rapm-2020-102084. PMID 34145074
- [Background] Koenen LR, Icenhour A, Forkmann K, Pasler A, Theysohn N, Forsting M, Bingel U, Elsenbruch S. Greater fear of visceral pain contributes to differences between visceral and somatic pain in healthy women. Pain. 2017 Aug;158(8):1599-1608. doi: 10.1097/j.pain.0000000000000924. PMID 28426553
- [Background] Rutherford D, Massie EM, Worsley C, Wilson MS. Intraperitoneal local anaesthetic instillation versus no intraperitoneal local anaesthetic instillation for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD007337. doi: 10.1002/14651858.CD007337.pub4. PMID 34693999
- [Background] Yong L, Guang B. Intraperitoneal ropivacaine instillation versus no intraperitoneal ropivacaine instillation for laparoscopic cholecystectomy: A systematic review and meta-analysis. Int J Surg. 2017 Aug;44:229-243. doi: 10.1016/j.ijsu.2017.06.043. Epub 2017 Jun 30. PMID 28669869
- [Background] Kang H, Kim BG. Intraperitoneal ropivacaine for effective pain relief after laparoscopic appendectomy: a prospective, randomized, double-blind, placebo-controlled study. J Int Med Res. 2010 May-Jun;38(3):821-32. doi: 10.1177/147323001003800309. PMID 20819419
- [Background] Ruiz-Tovar J, Gonzalez J, Garcia A, Cruz C, Rivas S, Jimenez M, Ferrigni C, Duran M. Intraperitoneal Ropivacaine Irrigation in Patients Undergoing Bariatric Surgery: a Prospective Randomized Clinical Trial. Obes Surg. 2016 Nov;26(11):2616-2621. doi: 10.1007/s11695-016-2142-z. PMID 27007272
- [Background] Gebhart GF, Bielefeldt K. Physiology of Visceral Pain. Compr Physiol. 2016 Sep 15;6(4):1609-1633. doi: 10.1002/cphy.c150049. PMID 27783853
- [Background] Kahokehr A, Sammour T, Zargar Shoshtari K, Taylor M, Hill AG. Intraperitoneal local anesthetic improves recovery after colon resection: a double-blinded randomized controlled trial. Ann Surg. 2011 Jul;254(1):28-38. doi: 10.1097/SLA.0b013e318221f0cf. PMID 21670611
- [Background] Schipper IE, Schouten M, Yalcin T, Algie GD, Damen SL, Smeenk RM, Schouten R. The Use of Intraperitoneal Bupivacaine in Laparoscopic Roux-en-Y Gastric Bypass: a Double-blind, Randomized Controlled Trial. Obes Surg. 2019 Oct;29(10):3118-3124. doi: 10.1007/s11695-019-03982-6. PMID 31201692
- [Background] Sparreboom CL, Wu Z, Dereci A, Boersema GS, Menon AG, Ji J, Kleinrensink GJ, Lange JF. Cytokines as Early Markers of Colorectal Anastomotic Leakage: A Systematic Review and Meta-Analysis. Gastroenterol Res Pract. 2016;2016:3786418. doi: 10.1155/2016/3786418. Epub 2016 Mar 9. PMID 27051416
- [Background] Wiik H, Karttunen R, Haukipuro K, Syrjala H. Maximal local and minimal systemic cytokine response to colorectal surgery: the influence of perioperative filgrastim. Cytokine. 2001 May 7;14(3):188-92. doi: 10.1006/cyto.2001.0870. PMID 11396998
- [Background] Zarbock A, Ley K. Neutrophil adhesion and activation under flow. Microcirculation. 2009 Jan;16(1):31-42. doi: 10.1080/10739680802350104. PMID 19037827
- [Background] Malsch P, Andratsch M, Vogl C, Link AS, Alzheimer C, Brierley SM, Hughes PA, Kress M. Deletion of interleukin-6 signal transducer gp130 in small sensory neurons attenuates mechanonociception and down-regulates TRPA1 expression. J Neurosci. 2014 Jul 23;34(30):9845-56. doi: 10.1523/JNEUROSCI.5161-13.2014. PMID 25057188
- [Background] Fang D, Kong LY, Cai J, Li S, Liu XD, Han JS, Xing GG. Interleukin-6-mediated functional upregulation of TRPV1 receptors in dorsal root ganglion neurons through the activation of JAK/PI3K signaling pathway: roles in the development of bone cancer pain in a rat model. Pain. 2015 Jun;156(6):1124-1144. doi: 10.1097/j.pain.0000000000000158. PMID 25775359
- [Background] Gudes S, Barkai O, Caspi Y, Katz B, Lev S, Binshtok AM. The role of slow and persistent TTX-resistant sodium currents in acute tumor necrosis factor-alpha-mediated increase in nociceptors excitability. J Neurophysiol. 2015 Jan 15;113(2):601-19. doi: 10.1152/jn.00652.2014. Epub 2014 Oct 29. PMID 25355965